CLINICAL TRIAL: NCT04789967
Title: The Effects of Imagery Treatments vs Progressive Muscle Relaxation Therapy in Terms of Clinical, Psychological and Physiological Aspects Among Patients With Functional Abdominal Bloating
Brief Title: Effects of Imagery Therapy vs Progressive Muscle Relaxation Therapy on Patients With Functional Abdominal Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Vincent Tee Wei Shen, Principle Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: USM/JEPeM/20110562
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Guided Imagery; Progressive Muscle Relaxation; Relaxation Techniques; Psychotherapy; Hypnosis; Sports Psychology; Bloating; Gastrointestinal Disease; Distention
MeSH Terms: conditions — Gastrointestinal Diseases; Dilatation, Pathologic | interventions — Imagery, Psychotherapy; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Imagery (GI) (Active Comparator): A 8 minute audio that focuses on evoking mental images in reducing the abdominal bloating sensation in patients
  Interventions: Behavioral: Guided Imagery
- Progressive Muscle Relaxation (PMR) (Active Comparator): A 8 minute audio that focuses on contracting certain muscle groups and relaxing it progressively in reducing the abdominal bloating sensation in patients
  Interventions: Behavioral: Progressive Muscle Relaxation
- Audiobook (Placebo Comparator): A 8 minute audio that focuses on providing educational information regarding functional gastrointestinal disorders and related knowledge.
  Interventions: Other: Educational Audiobook

INTERVENTIONS:
Behavioral: Guided Imagery — Individualized Guided Imagery (GI) technique, an alternative type of relaxation therapy. The content of GI usually includes scenery, places or any image projected to the mind. By using information generated, participants are guided to create a place in their mind using their senses of touch, sound, smell, sight and taste.
  Other Names: Imagery (Psychotherapy); Imagery, Guided; Psychotherapy Imagery; Imagery Psychotherapy
  Arms: Guided Imagery (GI)
Behavioral: Progressive Muscle Relaxation — Progressive muscle relaxation (PMR) therapy works by progressively relaxing and tensing the muscle groups throughout the entire body. Each muscle group will be tensed for about 5 seconds. If there's any pain or discomfort at any of the targeted areas, participants were told to omit that particular step. Constant purposeful deep breathing was instructed throughout the session especially in between changes of muscle.
  Other Names: Progressive Relaxation
  Arms: Progressive Muscle Relaxation (PMR)
Other: Educational Audiobook — Participants in the control group will receive an audiobook that targets to educate patients regarding gut-brain disorders, functional gastrointestinal disorders, causes of functional abdominal bloating, and treatment modalities available. Relaxing musical background will be added to facilitate the delivery.
  Arms: Audiobook

SUMMARY:
65% of the general population reported experiencing moderate to severe bloating symptoms. Bloating could be disturbing to patients and frustrating to the physicians as an effective treatment is still lacking. Guided Imagery (GI) involves the structured visualisation of mental images with somatic sensory; whereas Progressive Muscle Relaxation (PMR) focuses on tightening and relaxing the body's specific muscle groups. The development and validation of GI or PMR interventions to treat patients with functional abdominal bloating are relatively novel.

DETAILED DESCRIPTION:
The baseline variables of the patient would be obtained at the outpatient Gastrointestinal Medical clinic. A thorough general clinical interview that encompasses medical and psychological history, discussion of the nature and severity of the current symptoms, and review of past treatments and conclusions of any medical evaluation and tests. This is to make sure that the patients have been comprehensively evaluated medically and to rule out other causes of abdominal bloating before reaching a firm diagnosis of functional abdominal bloating as suggested in ROME IV Criteria. Questionnaires will be given out and patients were asked to fill it up on the spot. Electrical activity and abdominal circumference would be measured at an enclosed space with appropriate privacy and accompanied by a chaperone.

ELIGIBILITY:
Inclusion Criteria:

* Participants with abdominal bloating as determined using the Malay version Rome III criteria which was validated and translated by past researchers (Lee et al, 2012) and/or patients who were suggested by clinicians.
* Participants must be 18 years and above, and of either gender.
* Participants are able to read, write, or understand the Malay language.

Exclusion Criteria:

* Patients with abdominal bloating due to organic disorder
* Patients with recent abdominal surgeries (within 3 months) or previous major abdominal surgeries
* Patients with major neurological and psychological disorders including stroke, schizophrenia, major depression.
* Patients with medical history which may be the red flag for other FGIDs and organic disorders .
* Patients who are on psychotropic medications or psychotherapy which may confound outcome of imagery of sham intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Symptoms severity | 1 month
  Measured using the Malay version of Bloating Severity Questionnaire (BSQ-M). It consists of two components: five-item Sev24 and seven-item SevGen. The responses were in a multiple-choice answer format on different degrees of effect towards individuals on the basis of intensity, frequency and severity (less severe to more severe; range 1 to 4,5,6,7 or 8 varied by items). Higher scores in BSQ indicate worse severity.

SECONDARY OUTCOMES:
Health belief | 1 month
  Measured using the Malay-Language Health of Bloating (HB-Bloat) Scale. The questionnaire consists of 12 items and 3 domains: attitude (3 items), subjective norm (5 items), perceived control towards self-management (4 items). All responses were measured on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree).
Health seeking Intention | 1 month
  Measured using Health Seeking Intention for Abdominal Bloating Scale. It is a 5 point Likert scale that consists of 1 domain and 1 item. 1 indicates "strongly diagree" while 5 indicates "strongly agree"
Health promoting behavior | 1 month
  Measured using Health Promoting Behavior Scale of Abdominal Bloating. The questionnaire consists of 4 domains and 15 items. The questionnaire is a 5 point Likert scales, whereby 1 is considered strongly disagree and 5 is considered strongly agree.
Anxiety | 1 month
  Measured using the Malay version of Hospital Anxiety and Depression Scale (HADS). It comprises of 14 items, seven of which is related to anxiety symptoms. Each item is coded from 0 to 3. The scores for anxiety and depression can therefore vary from 0 to 21, depending on the presence and severity of the symptoms. A score between 0 and 7 does not indicate the presence of the symptoms of anxiety; a score between 8 and 10 indicates the presence of a moderate symptom; a score of 11 and above indicates a significant number of symptoms of anxiety corresponding to confirmed cases.
Depression | 1 month
  Measured using the Malay version of Hospital Anxiety and Depression Scale (HADS). It comprises of 14 items, seven of which is related to anxiety symptoms. Each item is coded from 0 to 3. The scores for anxiety and depression can therefore vary from 0 to 21, depending on the presence and severity of the symptoms. A score between 0 and 7 does not indicate the presence of the symptoms of anxiety; a score between 8 and 10 indicates the presence of a moderate symptom; a score of 11 and above indicates a significant number of symptoms of anxiety corresponding to confirmed cases.
Abdominal circumference | 1 month
  Using a non-stretch metric tape
Electrical activity | 1 month
  Measured using the Megawin ME6000 Electromyograph
Quality of life for patients with abdominal bloating | 1 month
  Measured using the Malay version of Bloating Quality of Life (BLQoL-M) Questionnaires. The responses for BLQoL were in a 7-point Likert scale on different degrees of impact towards individual ranging from 1 = "never/not related to me" to 7 = "always". Higher scores in BLQoL indicate higher impact towards QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Tee, MD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No